CLINICAL TRIAL: NCT03646916
Title: Effect of Pre-Operative Dexamethasone Dose on the Post-Operative Management of Blood Sugar in Diabetic Patients
Brief Title: Intraoperative Dexamethasone and Its Effect on Hyperglycemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Tarik Wasfie, MD, Principal Investigator, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GRMC160010
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone; Other: No dexamethasone
- Non-treatment (No Intervention)

INTERVENTIONS:
Drug: Dexamethasone — Gluco-corticosteroid
  Arms: Dexamethasone
Other: No dexamethasone — Nothing
  Arms: Dexamethasone

SUMMARY:
To study the effect of intra-operative dexamethasone on the management of post-operative blood sugar in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* documented history of Type I or Type II Diabetes Mellitus
* scheduled for surgery that requires patients to be admitted for at least 24 hours post-surgery

Exclusion Criteria:

* Patients on steroid therapy
* Pregnant women
* Patients at low risk for nausea/vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative blood sugar | 24 hour Post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States